CLINICAL TRIAL: NCT01533350
Title: Receptivity Assessment of Homogeneous Endometrium in Late Follicle Phase of Infertile Women With Natural Cycles
Brief Title: Receptivity Assessment of Homogeneous Endometrium in Late Follicle Phase
Status: Completed | Type: Observational
Sponsor: Shen-Zhen City Maternity and Child Healthcare Hospital (Other)
Responsible Party: Principal Investigator, Wen-Jie Zhu, Clinical Professor, Shen-Zhen City Maternity and Child Healthcare Hospital
Other Study IDs: 201002089
Record Dates: First submitted 2012-02-03; First posted 2012-02-15 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Infertile
Keywords: Ultrasonography; late follicle phase; homogeneous endometrium; receptivity; biochemical factor; ultrastructure; endometrial echo pattern
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The specimen was divided into three parts after washing with sterilized saline, and one was ﬁxed by 2.5% glutaraldehyde solution immediately ，then coated with palladium gold for electron microscopic examination;one was fixed by 2.5% glutaraldehyde arsenate ,then embedded in Epon for transmission electron microscopy ; one was ﬁxed by 4% formalin, then embedded in parafﬁn for immunohistochemical analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- group1: women with a ultrasonographic homogeneous echo endometrium in the late follicle phase
- group2: women with a ultrasonographic " triple-line" endometrium in the late follicle phase

SUMMARY:
Twenty eight infertile women undergoing ultrasonographic endometrial assessment in the late follicle phase, fourteen of them with homogeneous echo endometrium (group 1) and other fourteen with trilaminar endometrium (group 2), were included from our Department. The endometrial tissues were collected and Four biomarkers for endometrial receptivity and ultrastructure were assessed before and 6-7 days after ovulation.

DETAILED DESCRIPTION:
Subjects Twenty eight apparently healthy women, fourteen of them with a ultrasonographic homogeneous echo(group 1) and other fourteen with a " triple-line"(group 2) endometrium in the late follicle phase, were involved in our Department for the study between September 2010 and November 2011. The included criteria for both groups of women were ≤40 years of age, with a regular menstrual cycles (25-35 days), without use of an intrauterine devices or oral contraceptive at least 3 months before the study. Exclusion criteria were women with polycystic ovarian syndrome (PCOS), endometriosis, premature ovarian failure (POF) and an abortion within 1 year or a history of pelvic inflammatory disease. The mean age of the women were 31.9±3.7 years ( range, 26-39 years). The mean body mass index was 20.96±2.46 kg/m2 (range, 17.58-26.04 kg/m2).With a regular menstrual cycle (25-35days) and 2-11 years infertile history, all subjects had signed the proper consent forms. The study was approved by our Institutional Ethics committee.

Ovulation monitoring The women were followed for one cycle by obtaining blood samples and urine samples. The ovulation was monitored with vaginal ultrasonography (aloka-1000, UST-985, 5 MHz transvaginal probe, aloka Co. Ltd, Tokyo, Japan). The thickness of two endometrial layers was measured. The endometrial pattern was assessed according to the classification proposed by Gonen and Casper as follows: an endometrium that was entirely homogeneously hyperechoic without a central echogenic line was considered as a homogeneous echo pattern and triple-line pattern consisted of a central hyperechoic line surrounded by two hypoechoic layers. The growth of follicles, ovulation and the development of corpus luteum were monitored by using two-plane scans. Participants identified the day of the LH surge by testing the morning urine (David ovulation test, Rubio Biotech Co. Ltd., Shantou, China). The day of the LH surge was determined in urine samples when LH surge reached its highest value on which the blood samples were collected as well. The cycle day referred to the first day of menstrual bleeding. Women who have normal ovulatory cycles with intervals of 25-35 days are expected to ovulate on day 11 at the earliest and day 21at the latest. The peripheral blood samples were obtained by vein puncture on the day of the LH surge and 6-7 days after ovulation. Blood was separated by centrifugation within 1 hour, and the serum was stored at -20℃ until the concentrations of LH, FSH, estradiol (E2) and progesterone were assayed.

Endometrial biopsy Two endometrial biopsies were performed during a single menstrual cycle in each subject. The early biopsy was performed on the pre-ovulatory day (late follicle phase) and the endometrial tissues were collected from the anterior wall of the uterine cavity. Whereas the late biopsy was performed on ovulation day +7 (midluteal phase or implantation widow phase), and the endometrial sample was collected from the posterior wall of the uterine cavity with or without dilatation of the cervix by using an endometrial curette (#4164 prebet, Genetics, pommel, Belgium). Each sample was divided into three pieces and immediately fixed. Samples for scanning electron microscopy for fixed in a solution containing 2.5% (wt/vol) glutaraldehyde, 0.5% paraformaldehyde, 0.1 mol/L of sucrose, 0.1 mol/L of sodiumcacodylate, and 3 mmol/L of calciumchloride (pH, 7.4). Samples for immunohistochemistry were fixed in 4% formalin . Samples for transmission electron microscopy was fixed by 2.5% glutaraldehyde arsenate ;

Scanning electron microscopy Samples were washed twice in a buffer containing 0.15 mol/L of sodiumcacodylate and 3 mmol/L of calcium chloride (PH, 7.4) and once in distilled water. The specimens were dehydrated first in increasing concentrations of ethanol (70%,95%,and 99.5%) and then in acetone; they were dried in a critical-point dryer by using carbon dioxide. The specimens were mounted, coated with platinum, and examined by using a scanning electron microscope ( S-3000N, Hitachi, Tokyo, Japan). The developmental phase of the pinopode were classified. Because the pinopodes on the endometrial surface do not develop at exactly the same time the pinopodes were not evenly distributed over the endometrial surface, thus, in our study, we examined five fields each biopsy sample and analyzed the development and distribution of pinopodes. The morphology evaluation was defined as: no pinopodes,developing pinopodes,fully developed pinopodes and regressing pinopodes. The semi-quantitative evaluation was defined as following:- (0%), + (﹤20%), ++ (20-50%) and +++(>50%).

Immunohistochemistry 56 biopsy samples of 28 patients were used for immunohistochemical analysis. For LIF, integrin αv, VEGF and MMP-9 studies 4 um paraffin-embedded sections were deparaffinized 20 min in acetone at 70℃. Endogenous peroxidase was blocked with 3% H2O2 for 10 min. Antigen retrieval was boiling by heating for 5 min in 0.01 M citrate buffer at pH 6.0,and then the sections were incubated overnight at 4℃ with the specific antibodies which were diluted at 1:50. The antibodies used in this study were polyclonal antibodies (PAB) LIF, integrin αv, VEGF and MMP-9 (BA 1239, BA0957,BA0407 and BA0573, Booster Co Ltd, Wuhan, China). The sections were rinsed in phosphate-buffered saline (PBS), blocked with 10% normal goat serum for 30 min and then incubated with goat anti-rabbit biotinylated immunoglobulins (IgG)(SV0002, Booster Co Ltd, Wuhan, China) at 37℃ for 30 min. For integrin β3 study, the sections were incubated with 3% hydrogen peroxide for 10 min after hot repair of antigen by boiling at 95℃ of 0.01M citrate buffer(pH6.0), then incubated with polyclonal antibodies integrin β3 (sc-6626, santa, USA) diluted at 1:100 overnight at 4℃. Polymer Helper (PV-9003, Zhong-Shang Co Ltd, Beijing, China) was added at room temperature and with a interval of 20 min, Poly Peroxidase-anti-goat IgG (PV-9003, Zhong-Shang Co Ltd, Beijing, China) was added. The slides were then washed in PBS and colored by 3,3-diaminobenzidine in H2O2 (DAB, vitrogen, California, USA). The sections were finally washed in water. In every case a negative control was performed by omission of incubation with the primary specific antibody. The reactivity of each polyclonal antibody with endometrial glands and surface epithelium, stromal cells was assessed. Staining was evaluated semiquantitatively by using a grading system. Staining intensity and the number of stained cells were graded on a scale of 0=no staining, +/- = few stained cells, + = faint staining, ++ = moderate staining, and +++ = strong staining. The formula of H-score=ΣPi(i+1) was used to calculation. One observer who was blinded to identify of the slides performed all the assessments. After completion of the study, the same observer reexamined the slides to ensure reproducibility of the semiquantitative assessment.

Transmission electron microscopy Specimens for transmission electron microscopy were fixed in 2.5% glutaraldehyde in PBS (pH 7.4) and post-fixed in 1% osmium tetroxide. After dehydration in a graded ethanol series, specimens were placed in propylene oxide and embedded in Epon, stained with uranyl acetate and lead citrate and examined in transmission electron microscope .

Statistical Analysis The Statistics Package for Social Science (SPSS 13.0; SPSS Inc., Chicago, IL) was used for statistical analyses. The mean±S.D was evaluated using analysis of student's t-test ,ranked data was analyzed with the Rank Sum Test (Mann-Whitney test) and qualitative data was analyzed with chi-square test . Statistical significance was set at P<0.05(two tailed).

ELIGIBILITY:
Inclusion Criteria:

* infertile
* ≤ 40 years of age
* regular menstrual cycles (25-35 days)
* without use of an intrauterine devices or oral contraceptive at least 3 months before the study.

Exclusion Criteria:

* polycystic ovarian syndrome (PCOS)
* endometriosis
* premature ovarian failure (POF)
* an abortion within 1 year
* pelvic inflammatory disease history

Ages: 26 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The mean age of the women were 31.9±3.7 years ( range, 26-39 years). The mean body mass index was 20.96±2.46 kg/m2 (range, 17.58-26.04 kg/m2).With a regular menstral cycle (25-35days) and 2-11 years infertile history, all subjects had signed the proper consent forms.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
vascular endothelial growth factor（VEGF) | 2 month
  The expression analyzed by Immunohistochemistry.The stainings were graded semiquantitatively and the H-score was calculated using the following equation: H-score =∑Pi (i + 1), where i = intensity of staining with a value of 1, 2 or 3 (weak,moderate or strong, respectively) and Pi is the percentage of stained epithelial cells for each intensity, varying from 0 to 100%.
pinopodes | 2month
  The specimens were mounted, coated with platinum, and examined by using a scanning electron microscope ( S-3000N, Hitachi, Tokyo, Japan). The pinopodes morphology evaluation was defined as: no pinopodes,developing pinopodes,fully developed pinopodes and regressing pinopodes. The semi-quantitative evaluation was defined as following:- (0%), + (<20%), ++ (20-50%) and +++(>50%).
Ultrastructure | 2 month
  Ultrastructure was observed by transmission electron microscopy
leukemia inhibitory factor(LIF) | 2 months
  The expression analyzed by Immunohistochemistry.The stainings were graded semiquantitatively and the H-score was calculated using the following equation: H-score =∑Pi (i + 1), where i = intensity of staining with a value of 1, 2 or 3 (weak,moderate or strong, respectively) and Pi is the percentage of stained epithelial cells for each intensity, varying from 0 to 100%.
integrin ɑvβ3 | 2 months
  The expression analyzed by Immunohistochemistry.The stainings were graded semiquantitatively and the H-score was calculated using the following equation: H-score =∑Pi (i + 1), where i = intensity of staining with a value of 1, 2 or 3 (weak,moderate or strong, respectively) and Pi is the percentage of stained epithelial cells for each intensity, varying from 0 to 100%.
matrix metalloproteinase-9(MM-9) | 2 months
  The expression analyzed by Immunohistochemistry.The stainings were graded semiquantitatively and the H-score was calculated using the following equation: H-score =∑Pi (i + 1), where i = intensity of staining with a value of 1, 2 or 3 (weak,moderate or strong, respectively) and Pi is the percentage of stained epithelial cells for each intensity, varying from 0 to 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jie Zhu, M.D, Study Chair — Shenzhen Maternity and Child Healthcare Hospital
Locations (1):
- Department of Reproductive Healthcare, Shen-Zhen Maternity and Child Healthcare Hospital, Shenzhen, Guangdong, China